CLINICAL TRIAL: NCT06496451
Title: Measurement of Frataxin mRNA in NHP and Human Biofluids in Patients With Friedreich's Ataxia
Brief Title: Measurement of Frataxin mRNA in Biofluids
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 202301923
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich's Ataxia; Frataxin
MeSH Terms: conditions — Friedreich Ataxia | interventions — Spinal Puncture; Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Friedreich ataxia: Adult patients with genetically proven Friedreich ataxia
  Interventions: Other: Spinal tap for CSF collection; Other: Venipuncture for blood sample

INTERVENTIONS:
Other: Spinal tap for CSF collection — A spinal tap will be done on you by your choice of bedside or in the "interventional radiology (IR) suite" in the Shands (Neuromedicine) hospital. This procedure will be done by trained technicians under medical supervision or the principal investigator. Local anesthesia will be used to numb the site of injection on your back. We plan to collect about 4 tablespoons of spinal fluid.
Other: Venipuncture for blood sample — a sample of blood (approximately 4-5 tablespoonfuls) will be collected

SUMMARY:
The purpose of this research study is to determine a way to measure frataxin messenger RNA (mRNA) in fluids such as blood and cerebrospinal fluid (CSF) from patients with Friedreich's ataxia (FRDA). The gene mutation in FRDA leads to low levels of the mRNA and then low levels of the protein frataxin that leads to the disease. Treatments being developed for FRDA have the ability increase these levels including in brain where it is needed. Currently, there is no accepted way to measure frataxin protein or the messenger RNA (from which the protein is made) in the spinal fluid that surrounds the brain. In our study, the investigators aim to measure frataxin mRNA in both the blood and CSF. The investigators will use our ability to isolate structures called exosomes from these fluids. Exosomes are tiny, microscopic sacs that are known to contain many important biological molecules, and the investigators are able to detect frataxin mRNA in CSF from patients with other illnesses and from non-diseased participants. The investigators believe that parallel studies of exosomes in blood and CSF from patients with FRDA can tell us as to whether the frataxin mRNA in the CSF or blood of FRDA patients can serve as a measure of frataxin production in the brain. With one participation visit the investigators will be able to study the relationship of frataxin mRNA levels in the participant's CSF and blood with measures of disease severity. If successful, this will provide an important tool to monitor treatments for FRDA that aim to increase frataxin production.

DETAILED DESCRIPTION:
Overview of the Study Participants will complete the study during 2 visits (visit 1 and 2). Visit 1 can be combined with a routine clinic visit for care or research but also may be done remotely via Zoom. During visit 1, the investigators will fully explain the study and obtain the participant's informed consent. For remote visits, a copy of the consent will be emailed to the participant before the visit and the study team will schedule a time to discuss the consent. The informed consent will be reviewed in detail with the participant, and they will have an opportunity to ask any questions before signing the document and agreeing to the study. In either case, once the participant agrees to the study after being fully informed, they will sign the consent document and a copy of it will be provided to them after the investigator signs it.

Once informed consent has been obtained, the participant will either schedule visit 1 or begin visit 1 that day. Visit 1 will last no more than 2 hours and will involve the collection of clinical data and the collection of a blood sample. The participant will be asked to obtain lab work before visit 2, these labs will be to test the participant's blood for its ability to clot well. This lab work will be reviewed before visit 2. Visit 2 will take no more than 4 hours and will involve the collection of spinal fluid. The participant will need to be accompanied by a driver at visit 2.

Description of Study Procedures

Blood Work prior to scheduled visit (~30 minutes)

• will need to go to one of the University of Florida Health's (UF Health's) local labs in Gainesville, Florida (FL) to have blood work done before the scheduled visit 2. This blood work will ensure that the participant meet the inclusion criteria before the spinal tap.

Overall health and safety assessment (~30 minutes)

* The participant's birthdate, gender, contact information, health history, current medications, and allergies will be obtained. The information will be stored in the participant's study file.
* If the participant is a woman of childbearing potential, a urine sample will be tested to see if they are pregnant. If the test is positive, the participant will not be able to continue in the study.
* The participant's FRDA DNA test from their medical record will be assessed and a copy placed in the research folder. No additional genetic testing will be performed.
* Measurements such as the participant's height, weight, blood pressure, pulse, respiratory rate, and temperature will be obtained.
* A general physical examination will be done by the study physician

Neurological examination, modified Friedreich Ataxia Rating Scale (mFARS), and blood sample (~30 minutes)

* The study physician will perform a neurological examination and use this to rate the participant's ataxia severity in the mFARS scale.
* This will include examining the participant's eye movements, speech, strength of their muscles, sensation, coordination in their arms and legs and ability to stand and walk among other things.
* The participant will be asked questions regarding their activities of daily living for a questionnaire called FRDA activities of daily living scale (FARS ADL).
* A blood sample of approximately 5-10 milliliters (or 1-2 teaspoonfuls) will be obtained.

Spinal Tap (~3 hours)

* About 15 milliliters or 1 tablespoon of cerebrospinal fluid (CSF) will be collected though a test called a spinal tap.
* The spinal tap will be performed in the interventional radiology suite at the Neuromuscular hospital via x-ray fluoroscopy.
* This procedure uses X-ray (fluoroscopy) to visualize their low back spine so that the spinal tap needle can be placed in the spinal sac in the participant's low back under visual guidance. This can minimize discomfort and can help increase the success of the procedure in one attempt.
* The participant will be given local anesthesia to numb the area before collection.
* The participant will be asked to relax while laying down following the procedure for 1 to 2 hours before leaving.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Friedreich ataxia (men and women) related to documented biallelic GAA expansion in the FXN gene
* Age over 18 years
* No contraindication to spinal tap including any coagulopathy or local infections
* Competent to provide informed consent

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Any uncontrolled medical illness that may increase the risk of spinal tap such as ongoing infection as determined by the investigators
* FRDA related to an expansion in one allele and a conventional mutation on the other
* Positive pregnancy screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with Friedreich ataxia (FRDA)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Measurement of Frataxin mRNA in human biofluids | One year from final collection date
  The study plans to measure frataxin mRNA in exosomes from blood and spinal fluid as a biomarker in Friedreich ataxia

CONTACTS AND LOCATIONS:
Overall Officials: S H Subramony, M.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT06496451/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT06496451/ICF_001.pdf